CLINICAL TRIAL: NCT02066753
Title: The Cardiac Effects of Prolonged Hypothermia After Cardiac Arrest
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TTH48AG
Record Dates: First submitted 2014-02-17; First posted 2014-02-19 (Estimated); Last update posted 2015-11-25 (Estimated); Status verified 2015-11

CONDITIONS: Cardiac Arrest; Hypothermia
Keywords: Cardiac arrest; Therapeutic Hypothermia; Cardioprotectiveness; Hemodynamics
MeSH Terms: conditions — Heart Arrest; Hypothermia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 24 hours mild therapeutic hypothermia (Active Comparator): The patient will be treated with mild therapeutic hypothermia for 24 hours after reaching the target temperature between 32-34°C.
  Interventions: Procedure: Mild therapeutic hypothermia
- 48 hours mild therapeutic hypothermia (Experimental): The patient will be treated with mild therapeutic hypothermia for 48 hours after reaching the target temperature between 32-34°C.
  Interventions: Procedure: Mild therapeutic hypothermia

INTERVENTIONS:
Procedure: Mild therapeutic hypothermia — Mild therapeutic hypothermia with a target temperature between 32-34°C.

SUMMARY:
This PhD study is a sub study in a randomized clinical controlled multicenter trial named "TTH48" (ClinicalTrials.gov Identifier: NCT01689077).

The TTH48 trial examines prolonged mild therapeutic hypothermia ("MTH") at 32-34°C in 24 versus 48 hours with the primary outcome Cerebral Performance Category after 6 month in comatose out-of-hospital cardiac arrest patients.

THE OVERALL AIM OF THIS PhD STUDY IS TO INVESTIGATE THE CARDIAC FUNCTION AND THE HEMODYNAMICS BY BIOCHEMICAL CARDIAC MARKERS, ECHOCARDIOGRAPHY, BY ANALYZING THE USAGE OF INOTROPES/VASOPRESSORS AND BY ANALYZING ECG DATA FOR ARRHYTHMIAS IN THE 24 VERSUS 48 HOURS MTH GROUPS.

DETAILED DESCRIPTION:
The PhD-study contains 3 sub studies:

* Study 1 estimates the extend of myocardial damage resulting from the primary arrest and from the reperfusion injuries: Area under the curve of cTnT and CK-MB as 12 repeated measurements and NT-proBNP as 4 measurements post arrest

  -Hypothesis: There is a statistically significantly greater release of the cardiac biomarkers cTnT and NT-proBNP quantified by the area under the curve in the 24 versus the 48 hours group in the intervention period from 24 to 72 hours.
* Study 2 investigates MTH´s influence on systolic and diastolic function by standard and Tissue Doppler (TDI) echocardiography after 24, 48 and 72 hours. The primary endpoint is mitral annular systolic velocity ("S´ max")

  -Primary hypothesis: There is statistically significant improvement in S' max from the time T24 to T72 in the 48 versus the 24 hours group.

  -Secondary hypothesis: There is statistically significantly better systolic function at T48 measured in terms of individual S' max-change in the 48 hours group (still hypothermic) versus the 24 hours group (reached normothermia).
* Study 3 investigates MTH´s influence on the need for vasopressor or inotrope and the duration of arrhythmias during the first 72 hours post arrest.

  * Primary hypothesis: There is a statistically significantly increased tendency of arrhythmias in the 48 versus the 24 hours group measured in the period from T0 to T72.
  * Secondary hypothesis: There is a statistically significantly reduced need for inotropes in the 48 versus the 24 hours group measured by cumulative vasopressor index in the period from T0 to T72.

ELIGIBILITY:
Inclusion Criteria:

1. Resuscitated after cardiac arrest outside hospital with suspected cardiac triggering cause (and stabile circulation for at least 20 minutes after return of spontaneous circulation,
2. Glasgow coma score < 8 and
3. Age ≥ 18 years and < 80 years.

Exclusion Criteria:

1. Cardiac arrest of suspected non-cardiac triggering cause (e.g. trauma, aortic dissection, massive bleeding, hypoxia or accidental hypothermia),
2. >60 minutes from cardiac arrest to ROSC,
3. Time from cardiac arrest until start of cooling >4 hours,
4. Terminal illness,
5. Coagulopathy (medical anticoagulation treatment including thrombolysis is not a contraindication),
6. Unwitnessed arrests with asystolia as presenting rhythm,
7. Pregnancy,
8. Persistent cardiogenic shock,
9. Systolic blood pressure <80 mmHg despite vasoactive treatment and intra-aortic balloon pump
10. CPC 3-4 before the cardiac arrest,
11. Suspected/confirmed acute intra cerebral hemorrhage or stroke,
12. Acute CABG or other operation in connection with performing CPR,
13. Lack of consent from the relatives,
14. Lack of consent from the GP and
15. Lack of consent from the patient if he/she wakes up and is relevant.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-02; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Area under the curve cTnT | In the intervention period from 24 to 72 hours
  Allocated sub study 1
Mitral annular systolic velocity | After 24 hours, 48 hours and 72 hours
  Allocated sub study 2
Duration of arrhythmias | From target temperature (32-34°C) has been reached until 72 hours after
  Allocated sub study 3
Cumulative vasopressor index | From target temperature (32-34°C) has been reached until 72 hours after
  Allocated sub study 3

SECONDARY OUTCOMES:
Area under the curve NT-proBNP | In the intervention period from 24 to 72 hours
  Allocated sub study 1

CONTACTS AND LOCATIONS:
Overall Officials: Anders Grejs, MD, Principal Investigator — Research Center of Emergency Medicine and Department of Anesthesiology and Intensive Care Medicine, Aarhus University Hospital, Skejby, Denmark
Locations (2):
- Department of Anesthesiology and Intensive Care Medicine, Aarhus University Hospital, Skejby, Aarhus N, Central Jutland, Denmark
- Research Center of Emergency Medicine and Department of Anesthesiology and Intensive Care Medicine, Stavanger University Hospital, Stavanger, Norway

REFERENCES:
- [Derived] Jensen TH, Juhl-Olsen P, Nielsen BRR, Heiberg J, Duez CHV, Jeppesen AN, Frederiksen CA, Kirkegaard H, Grejs AM. Echocardiographic parameters during prolonged targeted temperature Management in out-of-hospital Cardiac Arrest Survivors to predict neurological outcome - a post-hoc analysis of the TTH48 trial. Scand J Trauma Resusc Emerg Med. 2021 Feb 19;29(1):37. doi: 10.1186/s13049-021-00849-7. PMID 33608045
- [Derived] Grejs AM, Nielsen BRR, Juhl-Olsen P, Gjedsted J, Sloth E, Heiberg J, Frederiksen CA, Jeppesen AN, Duez CHV, Hamre PD, Soreide E, Kirkegaard H. Effect of prolonged targeted temperature management on left ventricular myocardial function after out-of-hospital cardiac arrest - A randomised, controlled trial. Resuscitation. 2017 Jun;115:23-31. doi: 10.1016/j.resuscitation.2017.03.021. Epub 2017 Apr 2. PMID 28377297